CLINICAL TRIAL: NCT00043355
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II Study of Safety and Efficacy of Inhaled Interferon Gamma-1b With Antimycobacterials in Previously Treated or Mod-to-Sev Pulmonary Mycobacterium Avium Complex Infection
Brief Title: Safety and Efficacy of Inhaled Interferon Gamma-1b in Pulmonary MAC Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIMAC-001
Record Dates: First submitted 2002-08-07; First posted 2002-08-12 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Lung Infection
Keywords: pulmonary; mycobacterium avium complex infection; MAC; nontuberculous; mycobacteria; lung
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; Mycobacterium Infections | interventions — interferon gamma-1b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: interferon gamma-1b — 500 mcg, oral, three times weekly

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of inhaled Interferon gamma-1b (IFN-g 1b), when administered for 48 weeks and in combination with oral antibiotics which may be administered for up to 72 weeks for the treatment of a lung infection caused by a bacterium called Mycobacterium avium complex .

FDA has not approved Interferon gamma-1b for use in patients with MAC infection of the lungs, which is the purpose of this study.Interferon gamma-1b and similar proteins play important roles in establishing and maintaining protective immune responses against a variety of microorganisms.

DETAILED DESCRIPTION:
Laboratory research has shown that a mouse form of interferon gamma is effective in treating mice with infections caused by bacteria similar to MAC as well as MAC infection.

ELIGIBILITY:
Male and female patients, 18 years of age or older, with bacteriologically and radiographically confirmed pulmonary MAC infection who have been treated for their infection for at least 6 months within the previous 2 years, as well as patients with moderate or severe pulmonary disease due to MAC, not previously treated for this infection. Patients with recurrent pulmonary MAC infection after previous successful treatment for pulmonary MAC disease are also eligible.

In addition, various laboratory testing must confirm conditions. Patients cannot be positive for HIV or have an extra-pulmonary (in general, outside of the lungs) infection of MAC. Other preconditions related to health or other conditions exist as factors for inclusion or exclusion from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-12; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
sustained culture conversion | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Porter, MD, Study Director — InterMune